CLINICAL TRIAL: NCT03600818
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Sarilumab in Patients With Polymyalgia Rheumatica
Brief Title: Evaluation of the Efficacy and Safety of Sarilumab in Patients With Polymyalgia Rheumatica
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Protracted recruitment timeline exacerbated by COVID-19 pandemic
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EFC15160; 2017-002989-42 (EudraCT Number); U1111-1201-0777 (Other: UTN)
Record Dates: First submitted 2018-07-17; First posted 2018-07-26 (Actual); Results first posted 2022-06-10 (Actual); Last update posted 2022-06-10 (Actual); Status verified 2022-05

CONDITIONS: Polymyalgia Rheumatica
MeSH Terms: conditions — Polymyalgia Rheumatica | interventions — sarilumab; Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo+52 Week Taper (Placebo Comparator): Participants received sarilumab-matching placebo as subcutaneous (SC) injection every 2 weeks (q2w) up to 52 weeks along with the combination of prednisone and/or prednisone-matching placebo according to the protocol-defined schedule. Participants received prednisone/prednisone-matching placebo tapering oral daily doses for 52 weeks.
  Interventions: Drug: Sarilumab-matching placebo; Drug: Prednisone; Drug: Prednisone-matching placebo
- Sarilumab 200mg q2w+14 Week Taper (Experimental): Participants received sarilumab 200 milligrams (mg) as SC injection q2w up to 52 weeks along with the combination of prednisone and/or prednisone-matching placebo according to the protocol-defined schedule. Participants received prednisone tapering oral daily doses during the first 14 weeks and prednisone-matching placebo from Week 14 up to Week 52.
  Interventions: Drug: Sarilumab SAR153191 (REGN88); Drug: Prednisone; Drug: Prednisone-matching placebo

INTERVENTIONS:
Drug: Sarilumab SAR153191 (REGN88) — Pharmaceutical form:solution for injection Route of administration: subcutaneous
  Arms: Sarilumab 200mg q2w+14 Week Taper
Drug: Sarilumab-matching placebo — Pharmaceutical form:solution for injection Route of administration: subcutaneous
  Arms: Placebo+52 Week Taper
Drug: Prednisone — Pharmaceutical form:over-encapsulated tablets Route of administration: oral administration
Drug: Prednisone-matching placebo — Pharmaceutical form:over-encapsulated tablets Route of administration: oral administration
Drug: Prednisone — Pharmaceutical form:tablets Route of administration: oral administration

SUMMARY:
Primary Objective:

To evaluate the efficacy of KEVZARA (sarilumab) in participants with polymyalgia rheumatica (PMR) as assessed by the proportion of participants with sustained remission for sarilumab with a shorter corticosteroid (CS) tapering regimen as compared to placebo with a longer CS tapering regimen.

Secondary Objectives:

* To demonstrate the efficacy of sarilumab in participants with PMR compared to placebo, in combination with a CS taper with regards to:
* Clinical responses (such as components of sustained remission, disease remission rates, time to first disease flare) over time.
* Cumulative CS (including prednisone) exposure.
* To assess the safety (including immunogenicity) and tolerability of sarilumab in participants with PMR.
* To measure sarilumab serum concentrations in participants with PMR.
* To assess the effect of sarilumab in reducing glucocorticoid toxicity as measured by the composite glucocorticoid toxicity index (GTI) questionnaire.

DETAILED DESCRIPTION:
Study duration per participant was approximative 62 weeks including up to a 4-week screening period, 52-week treatment period and 6-week follow-up period.

ELIGIBILITY:
Inclusion criteria :

* Diagnosis of PMR according to European League Against Rheumatism/American College of Rheumatology classification criteria.
* Participants must be on prednisone of at least 7.5 milligrams per day (mg/day) (or equivalent) and not exceeding 20 mg/day at screening and during the screening period.
* Participant was willing and able to take prednisone of 15 mg/day at randomization.
* Participants had a history of being treated for at least 8 weeks with prednisone (greater than or equal to [>=]10 mg/day or equivalent).
* Participants must have had at least one episode of unequivocal PMR flare while attempting to taper prednisone at a dose that was >= 7.5 mg/day (or equivalent) within the past 12 Weeks prior to screening:

  * Unequivocal symptoms of PMR flare included shoulder and/or hip girdle pain associated with inflammatory stiffness.
* Participants had erythrocyte sedimentation rate >=30 millimeters per hour (mm/hr) and/or C-reactive protein >=10 milligrams per liter (mg/L) associated with PMR disease activity within 12 weeks prior to screening.

Exclusion criteria:

* Diagnosis of giant cell arteritis (e.g., persistent or recurrent localized headache, temporal artery or scalp tenderness, jaw claudication, extremity claudication, blurry or loss of vision, symptoms of stroke).
* Diagnosis of active fibromyalgia.
* Concurrent rheumatoid arthritis or other inflammatory arthritis or other connective tissue diseases, such as but not limited to systemic lupus erythematosus, systemic sclerosis, vasculitis, myositis, mixed connective tissue disease, and ankylosing spondylitis.
* Concurrent diagnosis of rhabdomyolysis or neuropathic muscular diseases.
* Inadequately treated hypothyroidism.
* Organ transplant recipient.
* Therapeutic failure including inadequate response or intolerance, or contraindication, to biological interleukin-6 antagonist.
* Any prior (within the defined period below) or concurrent use of immunosuppressive therapies but not limited to any of the following:

  * Janus kinase inhibitor within 4 weeks of Baseline.
  * Alkylating agents including cyclophosphamide within 6 months of Baseline.
  * Cell-depletion agents (e.g., anti CD20) without evidence of recovery of B cells to Baseline level.
  * Tumor necrosis factor inhibitors within 2-8 weeks (etanercept within 2 weeks, infliximab, certolizumab, golimumab, or adalimumab within 8 weeks), or after at least 5 half-lives have elapsed, whichever was longer.
  * Abatacept within 8 weeks of Baseline.
  * Anakinra within 1 week of Baseline.
  * Cyclosporine, azathioprine or mycophenolate mofetil or leflunomide within 4 weeks of Baseline.
* Unstable methotrexate (MTX) dose and/or MTX dose greater than (>) 15 mg/week within 3 months of Baseline
* Concurrent use of systemic CS for conditions other than PMR.
* Pregnant or breastfeeding woman.
* Participants with active or untreated latent tuberculosis.
* Participants with history of invasive opportunistic infections.
* Participants with fever associated with infection or chronic, persistent or recurring infections required active treatment.
* Participants with uncontrolled diabetes mellitus.
* Participants with non-healed or healing skin ulcers.
* Participants who received any live, attenuated vaccine within 3 months of Baseline.
* Participants who were positive for hepatitis B, hepatitis C and/or human immunodeficiency virus.
* Participants with a history of active or recurrent herpes zoster.
* Participants with a history of or prior articular or prosthetic joint infection.
* Prior or current history of malignancy.
* Participants who have had surgery within 4 weeks of screening or planned surgery during study.
* Participants with a history of inflammatory bowel disease or severe diverticulitis or previous gastrointestinal perforation.

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2018-10-09 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-05-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (84):
- United States (10):
  - Investigational Site Number 8400003, Upland, California
  - Investigational Site Number 8400005, Denver, Colorado
  - Investigational Site Number 8400009, Stamford, Connecticut
  - Investigational Site Number 8400002, Boca Raton, Florida
  - Investigational Site Number 8400014, Iowa City, Iowa
  - Investigational Site Number 8400006, Boston, Massachusetts
  - Investigational Site Number 8400022, New York, New York
  - Investigational Site Number 8400011, Dallas, Texas
  - Investigational Site Number 8400025, Lufkin, Texas
  - Investigational Site Number 8400015, Spokane, Washington
- Argentina (4):
  - Investigational Site Number 0320001, Buenos Aires
  - Investigational Site Number 0320005, Buenos Aires
  - Investigational Site Number 0320002, Caba
  - Investigational Site Number 0320003, San Miguel de Tucumán
- Australia (4):
  - Investigational Site Number 0360003, Camberwell
  - Investigational Site Number 0360001, Kogarah
  - Investigational Site Number 0360002, Maroochydore
  - Investigational Site Number 0360004, Woodville South
- Belgium (2):
  - Investigational Site Number 0560003, Ghent
  - Investigational Site Number 0560001, Leuven
- Canada (5):
  - Investigational Site Number 1240007, Hamilton
  - Investigational Site Number 1240010, Montreal
  - Investigational Site Number 1240001, Rimouski
  - Investigational Site Number 1240005, Sherbrooke
  - Investigational Site Number 1240003, Trois-Rivières
- Investigational Site Number 2330001, Tallinn, Estonia
- France (9):
  - Investigational Site Number 2500005, Brest
  - Investigational Site Number 2500011, Caen
  - Investigational Site Number 2500015, Le Kremlin-Bicêtre
  - Investigational Site Number 2500010, Lille
  - Investigational Site Number 2500002, Montivilliers
  - Investigational Site Number 2500003, Montpellier
  - Investigational Site Number 2500004, Paris
  - Investigational Site Number 2500016, Pierre-Bénite
  - Investigational Site Number 2500014, Toulouse
- Germany (7):
  - Investigational Site Number 2760008, Bad Abbach
  - Investigational Site Number 2760009, Berlin
  - Investigational Site Number 2760001, Berlin
  - Investigational Site Number 2760002, Dresden
  - Investigational Site Number 2760003, Kirchheim unter Teck
  - Investigational Site Number 2760004, München
  - Investigational Site Number 2760007, Tübingen
- Investigational Site Number 3480001, Debrecen, Hungary
- Israel (5):
  - Investigational Site Number 3760001, Haifa
  - Investigational Site Number 3760004, Haifa
  - Investigational Site Number 3760003, Kfar Saba
  - Investigational Site Number 3760002, Petah Tikva
  - Investigational Site Number 3760005, Tel Litwinsky
- Italy (6):
  - Investigational Site Number 3800003, Milan
  - Investigational Site Number 3800001, Milan
  - Investigational Site Number 3800004, Pisa
  - Investigational Site Number 3800002, Reggio Emilia
  - Investigational Site Number 3800005, Rozzano
  - Investigational Site Number 3800008, Verona
- Japan (4):
  - Investigational Site Number 3920002, Fuchu-Shi
  - Investigational Site Number 3920003, Kamakura-Shi
  - Investigational Site Number 3920005, Kawachinagano-Shi
  - Investigational Site Number 3920001, Takasaki-Shi
- Netherlands (6):
  - Investigational Site Number 5280003, Alkmaar
  - Investigational Site Number 5280002, Almelo
  - Investigational Site Number 5280005, Leeuwarden
  - Investigational Site Number 5280004, Nijmegen
  - Investigational Site Number 5280008, Rotterdam
  - Investigational Site Number 5280007, The Hague
- Russia (5):
  - Investigational Site Number 6430002, Moscow
  - Investigational Site Number 6430001, Moscow
  - Investigational Site Number 6430003, Moscow
  - Investigational Site Number 6430004, Moscow
  - Investigational Site Number 6430008, Saint Petersburg
- Spain (7):
  - Investigational Site Number 7240004, A Coruña / Santiago de Compostela
  - Investigational Site Number 7240005, Badalona
  - Investigational Site Number 7240001, Getafe
  - Investigational Site Number 7240008, Granada
  - Investigational Site Number 7240002, Madrid
  - Investigational Site Number 7240006, Santander
  - Investigational Site Number 7240007, Valencia
- Switzerland (2):
  - Investigational Site Number 7560001, Bern
  - Investigational Site Number 7560002, Sankt Gallen
- United Kingdom (6):
  - Investigational Site Number 8260004, Gateshead
  - Investigational Site Number 8260003, Leeds
  - Investigational Site Number 8260009, Manchester
  - Investigational Site Number 8260007, Newport
  - Investigational Site Number 8260002, Plymouth
  - Investigational Site Number 8260001, Southend

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org
URL: https://vivli.org

REFERENCES:
- [Derived] Strand V, Msihid J, Sloane J, Nivens MC, Chao J, Giannelou A, Fiore S, Araujo L, Dasgupta B. Sarilumab in relapsing polymyalgia rheumatica: patient-reported outcomes from a phase 3, double-blind, randomised controlled trial. Lancet Rheumatol. 2025 Aug;7(8):e544-e553. doi: 10.1016/S2665-9913(25)00041-4. Epub 2025 Jun 19. PMID 40544861
- [Derived] Spiera RF, Unizony S, Warrington KJ, Sloane J, Giannelou A, Nivens MC, Akinlade B, Wong W, Bhore R, Lin Y, Buttgereit F, Devauchelle-Pensec V, Rubbert-Roth A, Yancopoulos GD, Marrache F, Patel N, Dasgupta B; SAPHYR Investigators. Sarilumab for Relapse of Polymyalgia Rheumatica during Glucocorticoid Taper. N Engl J Med. 2023 Oct 5;389(14):1263-1272. doi: 10.1056/NEJMoa2303452. PMID 37792612

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 78 active centers (randomized at least 1 participant) in 17 countries. A total of 196 participants were screened between 09 October 2018 and 19 March 2020, of whom 78 were screen failures. Screen failures were mainly due to not meeting inclusion criteria.
Pre-assignment Details: Participants were randomized to two treatment groups in a 1:1 ratio by interactive response technology. A total of 118 participants were enrolled and randomized in the study.
Period: Overall Study
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Started | 58 | 60
Safety Population (All randomized participants who received at least one dose or part of a dose of the study medication (IMP) analyzed according to the treatment they actually received.) | 58 | 59
Completed | 36 | 42
Not Completed | 22 | 18
Not completed — Adverse Event | 4 | 7
Not completed — Lack of Efficacy | 9 | 4
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Other-unspecified | 5 | 3
Not completed — Randomized and not treated | 0 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on randomized population.
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper | Total Title
Number analyzed (Participants) | 58 | 60 | 118
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.1 (8.5) | 68.8 (7.8) | 68.9 (8.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 45 | 82
  Male | 21 | 15 | 36
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 48 | 50 | 98
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 8 | 9 | 17

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Sustained Remission at Week 52
Description: Sustained remission was defined as meeting all of the following parameters: achievement of disease remission (defined as resolution of signs and symptoms of polymyalgia rheumatica [PMR], and normalization of C-reactive protein [CRP] {less than [<]10 milligrams per liter [mg/L]}) not later than Week 12, absence of disease flare (defined as recurrence of signs and symptoms attributable to active PMR plus an increase in corticosteroid [CS] dose due to PMR or elevation of erythrocyte sedimentation rate [ESR] attributable to active PMR plus an increase in CS dose due to PMR) from Week 12 through Week 52, sustained reduction of CRP (to <10 mg/L, with absence of successive elevations to greater than or equal to [>=]10 mg/L) from Week 12 through Week 52, and successful adherence to prednisone taper from Week 12 through Week 52.
Time Frame: At Week 52
Population: Analysis was performed on intent-to-treat (ITT) population that included all participants who were allocated to a randomized treatment group, and were analyzed according to the treatment group allocated by randomization.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58 | 60
percentage of participants | 10.3 | 28.3
Statistical Analysis 1: Comparison: Placebo+52 Week Taper vs Sarilumab 200mg q2w+14 Week Taper; Test type: Superiority; p = 0.0193, Fisher Exact — Threshold for significance at 0.05 level; Difference in percentage = 18.0, 95% CI 2-sided [4.15 to 31.82]

2. Secondary Outcome: Total Cumulative Corticosteroid Dose
Description: Cumulative dose of CS used for PMR disease was defined as the dose taken up to the end of treatment, including expected prednisone in tapering regimen per protocol, add-on prednisone, CS used in rescue therapy and the use of commercial prednisone (an excess of <=100 mg of prednisone during the study treatment period). The total cumulative CS dose was based on the total number of days with complete or partial intake, no imputation was done on missed tablets.
Time Frame: Up to Week 52
Population: Analysis was performed on ITT population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58 | 59
milligrams | 2235.8 (839.4) | 1039.5 (612.2)
Statistical Analysis 1: Comparison: Placebo+52 Week Taper vs Sarilumab 200mg q2w+14 Week Taper; A hierarchical testing procedure was used to control the overall type I error. If the primary endpoint reaches statistical significance then the secondary endpoint for total cumulative CS dose was tested next; Test type: Superiority; p < 0.0001, Wilcoxon rank-sum test — Threshold for significance at 0.05 level

3. Secondary Outcome: Number of Participants Who Achieved Disease Remission up to Week 12
Description: Disease remission was defined as resolution of signs and symptoms of PMR, and normalization of CRP (< 10 mg/L). The status of normalization of CRP (<10 mg/L) was determined based on the last two non-missing post-baseline CRP values measured up to Week 12. If at least one of the value was <10 mg/L, then it was considered as normalization of CRP. Participants who took rescue CS due to active PMR prior to Week 12 or who permanently withdrew from the study treatment prior to Week 12 were considered as not achieved disease remission by Week 12. During the initial 12 weeks of prednisone taper, treatment for one flare before Week 12 was permitted if it was successfully treated with a low dose (<=5 mg/day) prednisone add-on taper regimen (completed prior to Week 12) and provided that all other sustained remission parameters were met.
Time Frame: Up to Week 12
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58 | 60
Participants | 22 | 28

4. Secondary Outcome: Number of Participants With Absence of Disease Flare From Week 12 Through Week 52
Description: Disease flare was defined as either recurrence of signs and symptoms attributable to active PMR plus an increase in CS dose due to PMR, or elevation of ESR attributable to active PMR plus an increase in CS dose due to PMR.
Time Frame: From Week 12 Through Week 52
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58 | 60
Participants | 19 | 33

5. Secondary Outcome: Number of Participants With Sustained Reduction of CRP From Week 12 Through Week 52
Description: Normalization (sustained reduction) of CRP was defined as CRP levels <10 mg/L. If there were two or more consecutive visits with CRP >=10 mg/L, then it was categorized as no normalization of CRP.
Time Frame: From Week 12 through Week 52
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58 | 60
Participants | 26 | 40

6. Secondary Outcome: Number of Participants With Successful Adherence to the Prednisone Taper From Week 12 Through Week 52
Description: Successful adherence to the prednisone taper from Week 12 through Week 52 was defined as participants who did not take rescue therapy from Week 12 through Week 52 and any excess prednisone (beyond the per protocol CS tapering regimen) with a cumulative dose of <=100 mg (or equivalent), such as those employed to manage adverse event (AE) not related to PMR.
Time Frame: From Week 12 through Week 52
Population: Analysis was performed on ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58 | 60
Participants | 14 | 30

7. Secondary Outcome: Time to First Polymyalgia Rheumatica Flare After Clinical Remission up to Week 52
Description: Time to first PMR flare was defined as the duration (in days) from randomization to first PMR flare after clinical remission (defined as resolution of signs and symptoms and normalization of CRP [<10 mg/L]) and up to 52 weeks. Disease flare was defined as either the recurrence of signs or symptoms attributable to active plus an increase in CS dose due to PMR or elevation of ESR attributable to active PMR plus an increase in CS dose due to PMR. Kaplan-Meier method was used for the analysis. Participants who never achieved remission were censored at randomization day; and those who achieved clinical remission and never flared were censored at the end of treatment assessment date up to Week 52.
Time Frame: Up to Week 52
Population: Analysis was performed on ITT population.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58 | 60
days | 99.00 [1.000 to 154.000] | NA [93.000 to NA] — At Week 52 the cumulative incidence was less than 50% in the Kaplan-Meier plot. Hence, the upper limit of confidence interval and median value was not reached.

8. Secondary Outcome: Composite Glucocorticoid Toxicity Index (C-GTI): Cumulative Worsening Score (CWS) and Aggregate Improvement Score (AIS) at Week 52
Description: GTI assessed glucocorticoid (GC) related morbidity and GC-sparing ability of other therapies; composed of 2 components: C-GTI and Specific List. C-GTI contained 9 domains and Specific List contained of 23 items (11 domains), used as complementary tool to C-GTI. C-GTI score was sum of 9 domain-specific scores at each visit and Cumulative GTI score was sum of C-GTI scores across each visit. Two cumulative GTI scores: CWS and AIS at Week 52 are reported in this outcome measure. CWS assessed cumulative GC toxicity regardless of whether toxicity had lasting effects or was transient. AIS assessed new therapy effectiveness in decreasing any Baseline GC toxicity over time. Negative scores reflect improvement in CS toxicities present from Baseline. For CWS, composite score ranged from 0 to 439 and for AIS, composite score ranged from -346 to 439. For both CWS and AIS, minimum score implies least toxicity and maximum score implies most toxicity.
Time Frame: At Week 52
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 57 | 60
units on a scale
  CWS | 57.22 (6.678) | 52.32 (6.507)
  AIS | 2.57 (6.275) | -4.02 (6.115)

9. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Treatment-emergent Serious Adverse Events (TESAEs)
Description: An AE was defined as any untoward medical occurrence in a participant who received study drug and did not necessarily had to have a causal relationship with the treatment. Serious AEs (SAEs) were any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial or prolonged in-patient hospitalization, persistent or significant disability/incapacity, congenital anomaly/birth defect, or considered as medically important event. TEAEs were the AEs that developed or worsened or became serious during the TEAE period (defined as the time from the first dose of the investigational medicinal product (IMP) to the last dose of the IMP +60 days).
Time Frame: From first dose (i.e. Day 1) up to 60 days after last dose date of study drug (i.e. up to Week 60)
Population: Analysis was performed on safety population that included participants who had received at least one dose or part of a dose of IMP and were analyzed according to the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58 | 59
Participants
  Any TEAE | 49 | 56
  TESAE | 12 | 8

10. Secondary Outcome: Number of Participants With Potentially Clinically Significant Vital Signs Abnormalities During TEAE Period
Description: Criteria for potentially clinically significant vital sign abnormalities:
  Systolic Blood Pressure (SBP): <= 95 mmHg and decrease from baseline (DFB) more than or equal to (>=) 20 mmHg; >= 160 mmHg and increase from baseline (IFB) >= 20 mmHg
  Diastolic blood pressure (DBP): <=45 mmHg and DFB >=10 mmHg; >=110 mmHg and IFB >=10 mmHg.
  Heart Rate (HR): <= 50 beats per min (bpm) and DFB >=20 bpm; >=120 bpm and IFB >= 20 bpm
  Weight: >=5% DFB; >=5% IFB.
  TEAE period was defined as the time from the first dose of the IMP to the last dose of the IMP + 60 days.
Time Frame: From first dose (i.e., Day 1) up to 60 days after last dose date of study drug (i.e., up to Week 60)
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure and 'number analyzed' = participants with available data for each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58 | 58
Participants
  SBP <=95 mmHg and DFB >=20 mmHg | 0 | 2
  SBP >=160 mmHg and IFB >=20 mmHg | 4 | 5
  DBP <=45 mmHg and DFB >=10 mmHg | 1 | 0
  DBP >=110 mmHg and IFB >=10 mmHg | 1 | 1
  HR <=50 bpm and DFB >= 20 bpm | 1 | 0
  HR >=120 bpm and IFB >=20 bpm | 1 | 0
  Weight >=5% DFB: number analyzed (Participants) | 56 | 58
  Weight >=5% DFB | 2 | 5
  Weight >=5% IFB: number analyzed (Participants) | 56 | 58
  Weight >=5% IFB | 9 | 12

11. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities - Hematological Parameter
Description: Criteria for potentially clinically significant laboratory abnormalities included:
  Hemoglobin (Hb): <= 115 grams per liter (g/L) (Male [M]), <= 95 g/L (Female [F]); >= 185 g/L (M), >= 165 g/L (F); DFB >= 20 g/L .
  Hematocrit: <= 0.37 volume/volume (v/v) (M); <= 0.32 v/v (F); >= 0.55 v/v (M); >= 0.5 v/v (F).
  Erythrocytes: >=6 Tera/ liter (L).
  Platelets: < 100 Giga/L, >= 700 Giga/L.
  Leukocytes: < 3.0 Giga/L (Non-Black [NB]); < 2.0 Giga/L (Black [B]), >= 16.0 Giga/L.
  Neutrophils: < 1.5 Giga/L (NB); < 1.0 Giga/L (B).
  Lymphocytes: > 4.0 Giga/L.
  Monocytes: > 0.7 Giga/L.
  Basophils: > 0.1 Giga/L.
  Eosinophils: > 0.5 Giga/L or > upper limit of normal (ULN) (if ULN >= 0.5 Giga/L).
Time Frame: From first dose (i.e., Day 1) up to 60 days after last dose date of study drug (i.e., up to Week 60)
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 57 | 58
Participants
  Hb: <= 115 g/L (M), <= 95 g/L (F) | 1 | 1
  Hb: >=185 g/L(M), >=165 g/L(F) | 0 | 1
  Hb: DFB >=20 g/L | 3 | 2
  Hematocrit: <= 0.37 v/v(M); <=0.32 v/v(F) | 1 | 1
  Hematocrit: >=0.55 v/v(M); >=0.5 v/v(F) | 0 | 0
  Erythrocytes: >=6 Tera/L | 0 | 0
  Platelets: < 100 Giga/L | 0 | 2
  Platelets: >= 700 Giga/L | 0 | 0
  Leukocytes:<3.0Giga/L(NB);<2.0Giga/L(B) | 0 | 11
  Leukocytes: >= 16.0 Giga/L. | 1 | 1
  Neutrophils: < 1.5 Giga/L (NB); < 1.0 Giga/L (B). | 0 | 18
  Lymphocytes: > 4.0 Giga/L | 4 | 2
  Monocytes: > 0.7 Giga/L | 12 | 8
  Basophils: > 0.1 Giga/L. | 16 | 13
  Eosinophils:>0.5 Giga/L; >ULN (if ULN>=0.5Giga/L) | 2 | 2

12. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities - Metabolic Parameters
Description: Criteria for potentially clinically significant abnormalities:
  Glucose: <=3.9 millimoles (mmol)/L and < lower limit of normal (LLN); >=11.1 mmol/L (unfasted [unfas]); >=7 mmol/L (fasted [fas]).
  HbA1c: >8%.
  Cholesterol: >=7.74 mmol/L.
  Triglycerides: >=4.6 mmol/L.
  C Reactive Protein (CRP): >2 ULN or >10 mg/L (if ULN not provided).
Time Frame: From first dose (i.e., Day 1) up to 60 days after last dose date of study drug (i.e., up to Week 60)
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58 | 58
Participants
  Glucose: <=3.9 mmol/L and < LLN: number analyzed (Participants) | 56 | 57
  Glucose: <=3.9 mmol/L and < LLN | 1 | 2
  Glucose: >=11.1 mmol/L (unfas); >=7 mmol/L (fas): number analyzed (Participants) | 56 | 57
  Glucose: >=11.1 mmol/L (unfas); >=7 mmol/L (fas) | 14 | 5
  HbA1c: >8% | 4 | 2
  Cholesterol: >=7.74 mmol/L | 4 | 8
  Triglycerides: >=4.6 mmol/L | 1 | 3
  CRP: >2 ULN or >10 mg/L (if ULN not provided) | 37 | 13

13. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities - Renal Function
Description: Criteria for potentially clinically significant abnormalities:
  Creatinine: >=150 micromol/L (adults); >=30% change from baseline, >=100% change from baseline.
  Creatinine clearance: >=60 to <90 milliliters per minute (mL/min); >=30 to <60 mL/min ; >=15 to <30 mL/min; <15 mL/min.
  Blood urea nitrogen: >=17 mmol/L.
  Urate: <120 micromol/L; >408 micromol/L.
Time Frame: From first dose (i.e., Day 1) up to 60 days after last dose date of study drug (i.e., up to Week 60)
Population: Analysis was performed on safety population. Here, 'overall number of participants analyzed'= participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58 | 58
Participants
  Creatinine: >=150 micromol/L (adults) | 2 | 2
  Creatinine: >=30% change from baseline | 3 | 14
  Creatinine: >=100% change from baseline | 0 | 1
  Creatinine clearance: >=60 to <90 mL/min | 30 | 29
  Creatinine clearance: >=30 to <60 mL/min | 13 | 17
  Creatinine clearance: >=15 to <30 mL/min | 0 | 1
  Creatinine clearance: <15 mL/min | 0 | 0
  Blood urea nitrogen: >=17 mmol/L | 0 | 0
  Urate: <120 micromol/L | 0 | 0
  Urate: >408 micromol/L | 16 | 16

14. Secondary Outcome: Number of Participants With Potentially Clinically Significant Abnormalities - Liver Function
Description: Criteria for potentially clinically significant abnormalities:
  Albumin: <= 25 g/L.
  Alanine Aminotransferase (ALT): >3 ULN; >5 ULN; >10 ULN.
  Aspartate Aminotransferase (AST): >3 ULN; >5 ULN; >10 ULN; >20 ULN.
  Alkaline Phosphatase: >1.5 ULN.
  Bilirubin: >1.5 ULN; >2 ULN.
  ALT and Total Bilirubin: ALT > 3 ULN and Bilirubin > 2 ULN
Time Frame: From first dose (i.e., Day 1) up to 60 days after last dose date of study drug (i.e., up to Week 60)
Population: as for outcome 11
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58 | 58
Participants
  Albumin: <= 25 g/L | 0 | 0
  ALT: >3 ULN | 2 | 0
  ALT: >5 ULN | 1 | 0
  ALT: >10 ULN | 0 | 0
  AST: >3 ULN | 1 | 0
  AST: >5 ULN | 1 | 0
  AST: >10 ULN | 1 | 0
  AST: >20 ULN | 0 | 0
  Alkaline Phosphatase: >1.5 ULN | 1 | 0
  Bilirubin: >1.5 ULN | 1 | 1
  Bilirubin: >2 ULN | 0 | 0
  ALT > 3 ULN and Bilirubin > 2 ULN | 0 | 0

15. Secondary Outcome: Number of Participants With Treatment-emergent Antidrug Antibodies (ADA) Response
Description: ADA response categories: 1) Treatment-boosted ADA positive participant: Participant with a positive ADA assay response at Baseline and with at least a 4-fold increase in titer compared to Baseline during TEAE period. 2) Treatment-emergent ADA positive participant: Participant with non-positive assay (meaning negative or missing) response at Baseline but with a positive assay response during the TEAE period (defined as the time from the first dose of the IMP to the last dose of the IMP +60 days).
Time Frame: From first dose (i.e., Day 1) up to 60 days after last dose date of study drug (i.e., up to Week 60)
Population: Analysis was performed on ADA population which included participants who had received at least one dose or part of a dose of IMP and were analyzed according to the treatment actually received and had at least one post dose evaluable ADA sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 55 | 56
Participants
  Treatment-boosted ADA | 0 | 0
  Treatment-emergent ADA | 1 | 2

16. Secondary Outcome: Pharmacokinetics (PK): Serum Trough Concentration (Ctrough) of Sarilumab
Description: Ctrough was pre dose concentration of drug. Data for this outcome measure was not planned to be collected and analyzed for placebo arm (Placebo+52 Week Taper) as pre-specified in the protocol.
Time Frame: Pre-dose on Week 0 (Baseline), Week 2, 4, 12, 16, 24, and 52
Population: Analyzed on PK population: participants who had received at least one dose or part of a dose of IMP, were analyzed according to the treatment actually received and had at least 1 post-dose non-missing serum sarilumab concentration value. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 58
nanograms per milliliter (ng/mL)
  Baseline | 0.00 (0.00)
  Week 2: number analyzed (Participants) | 56
  Week 2 | 5209.02 (4357.37)
  Week 4: number analyzed (Participants) | 50
  Week 4 | 9259.25 (7668.95)
  Week 12: number analyzed (Participants) | 46
  Week 12 | 17494.20 (11146.33)
  Week 16: number analyzed (Participants) | 42
  Week 16 | 23082.86 (15878.92)
  Week 24: number analyzed (Participants) | 40
  Week 24 | 27289.75 (17927.73)
  Week 52: number analyzed (Participants) | 33
  Week 52 | 27604.95 (24880.13)

17. Secondary Outcome: Pharmacokinetics: Serum Drug Concentration of Sarilumab Post-dose at Week 24
Description: Serum concentrations of functional sarilumab were analyzed using validated enzyme linked immunosorbent assay.
Time Frame: Post-dose at Week 24
Population: Analysis was performed on PK population. Here, 'overall number of participants analyzed' = participants evaluable for this outcome measure. Data for this outcome measure was not planned to be collected and analyzed for placebo arm (Placebo+52 Week Taper) as pre-specified in the protocol.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sarilumab 200mg q2w+14 Week Taper
Number analyzed (Participants) | 26
ng/mL | 35757.69 (15353.96)

ADVERSE EVENTS:
Time Frame: From first dose (i.e., Day 1) of IMP to last dose date of IMP + 60 days (i.e., up to Week 60).
Description: Reported AEs were TEAEs that developed/worsened in grade or became serious during TEAE period (defined as the time from the first dose of the IMP to the last dose of the SC IMP + 60 days). Analysis was performed on safety population.
Arm/Group | Placebo+52 Week Taper | Sarilumab 200mg q2w+14 Week Taper
All-Cause Mortality (participants affected / at risk) | 0/58 | 0/59
Serious Adverse Events (participants affected / at risk) | 12/58 | 8/59
Other Adverse Events (participants affected / at risk) | 42/58 | 42/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+52 Week Taper (N=58) | Sarilumab 200mg q2w+14 Week Taper (N=59)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Covid-19 (Infections and infestations) | 2 (2) | 0 (0)
Covid-19 Pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Intervertebral Discitis (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Urinary Tract Infection Bacterial (Infections and infestations) | 0 (0) | 1 (1)
Femur Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine Aminotransferase Increased (Investigations) | 1 (1) | 0 (0)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar Spinal Stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Polymyalgia Rheumatica (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Erdheim-Chester Disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Aortic Intramural Haematoma (Vascular disorders) | 0 (0) | 1 (1)
Giant Cell Arteritis (Vascular disorders) | 1 (1) | 1 (1)
Hypertensive Emergency (Vascular disorders) | 1 (1) | 0 (0)
Orthostatic Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo+52 Week Taper (N=58) | Sarilumab 200mg q2w+14 Week Taper (N=59)
Increased Tendency To Bruise (Blood and lymphatic system disorders) | 4 (4) | 4 (4)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (4)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 7 (9)
Dry Eye (Eye disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 4 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 7 (7)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 (2) | 3 (3)
Fatigue (General disorders) | 0 (0) | 3 (3)
Injection Site Pruritus (General disorders) | 0 (0) | 3 (7)
Oedema Peripheral (General disorders) | 5 (5) | 3 (3)
Cystitis (Infections and infestations) | 3 (4) | 2 (2)
Gastroenteritis (Infections and infestations) | 3 (4) | 2 (2)
Influenza (Infections and infestations) | 4 (4) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (6) | 2 (2)
Upper Respiratory Tract Infection (Infections and infestations) | 5 (5) | 2 (2)
Accidental Overdose (Injury, poisoning and procedural complications) | 1 (1) | 3 (4)
Fall (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Limb Injury (Injury, poisoning and procedural complications) | 3 (3) | 0 (0)
Skin Laceration (Injury, poisoning and procedural complications) | 3 (5) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 9 (11)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (3) | 3 (4)
Bursitis (Musculoskeletal and connective tissue disorders) | 5 (5) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (6)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Rotator Cuff Syndrome (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Tendonitis (Musculoskeletal and connective tissue disorders) | 2 (2) | 3 (5)
Cognitive Disorder (Nervous system disorders) | 4 (4) | 4 (4)
Headache (Nervous system disorders) | 5 (5) | 1 (1)
Sciatica (Nervous system disorders) | 1 (2) | 3 (3)
Depression (Psychiatric disorders) | 6 (7) | 5 (5)
Insomnia (Psychiatric disorders) | 9 (9) | 6 (6)
Mania (Psychiatric disorders) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (4)
Skin Striae (Skin and subcutaneous tissue disorders) | 4 (4) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 6 (6)

LIMITATIONS AND CAVEATS:
Protracted recruitment timeline exacerbated by COVID-19 pandemic led to pre-mature termination of study, resulting in a change in the total expected number of participants and change in the statistical significance level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/18/NCT03600818/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-20): https://cdn.clinicaltrials.gov/large-docs/18/NCT03600818/SAP_001.pdf